CLINICAL TRIAL: NCT07035119
Title: Transcranial Magnetic Stimulation for Chronic Scrotal Content Pain
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00140222
Record Dates: First submitted 2025-04-07; First posted 2025-06-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Scrotal Pain
Keywords: Scrotal pain; testicular pain; Transcranial magnetic stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label (Experimental): Open label study. Participants will be screened by study staff for contraindications to TMS treatment. TMS will be delivered use the MagVenture TMS machine.
  Interventions: Other: Transcranial magnetic stimulation

INTERVENTIONS:
Other: Transcranial magnetic stimulation — Resting motor threshold will be established by first finding the area of the motor cortex associated with visible twitch of the right abductor pollicis brevis (APB). Parameter Estimation by Sequential Testing (PEST) will be conducted to quantify resting motor threshold using visible APB twitch. The left dorsolateral prefrontal cortex (DLPFC) will be located using the Beam F3 method and marked with a felt-tipped marker on the scalp. TMS will be delivered over left DLPFC at 110% of resting motor threshold at 10Hz (5-seconds-on; 10-seconds-off) for 15 minutes per session (3000 pulses), 3 sessions each day (30-minute rest in-between sessions), for 3 days (within 5 consecutive days; a total of 27,000 pulses).

SUMMARY:
The purpose of this study is to perform an open label feasibility trial of TMS for the treatment of chronic scrotal content pain.

DETAILED DESCRIPTION:
The purpose of this study is to perform an open label feasibility trial of TMS for the treatment of chronic scrotal content pain. Participants will be screened by study staff for contraindications to TMS treatment. TMS will be delivered use the MagVenture TMS machine. TMS will be delivered during 15 minutes per session, 3 sessions each day, for 3 days. A custom developed SMS text EMA system will be used to gather daily data on pain and functioning in study participants.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with chronic scrotal pain lasting for 6 or more months.
* Pain must be present 3 or more days of the week.

Exclusion Criteria:

* No new pain medications within the last 30 days.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male (biological), with testis
Enrollment: 50 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported pain score on SMS text EMA system | baseline, and post intervention (0 days, 1 week, 2 weeks, 1 month, 3 months, 6 months)
  A custom developed SMS text EMA system will be used to gather daily data on pain

SECONDARY OUTCOMES:
Patient reported post procedure quality of life as measured on an SMS text EMA system | baseline, and post intervention (0 days, 1 week, 2 weeks, 1 month, 3 months, 6 months)
  A custom developed SMS text EMA system will be used to gather daily data on pain
Progression to other treatments | Within 6 months after completion
  Progression to other medical or surgical treatments

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Brockardt, Ph.D., Study Director — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Based on internal IRB submission, IPD will not be shared

REFERENCES:
- [Background] O'Connell NE, Wand BM, Marston L, Spencer S, Desouza LH. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2014 Apr 11;(4):CD008208. doi: 10.1002/14651858.CD008208.pub3. PMID 24729198
- [Background] Hamid P, Malik BH, Hussain ML. Noninvasive Transcranial Magnetic Stimulation (TMS) in Chronic Refractory Pain: A Systematic Review. Cureus. 2019 Oct 29;11(10):e6019. doi: 10.7759/cureus.6019. PMID 31824787
- [Background] Parekattil SJ, Ergun O, Gudeloglu A. Management of Chronic Orchialgia: Challenges and Solutions - The Current Standard of Care. Res Rep Urol. 2020 Jul 2;12:199-210. doi: 10.2147/RRU.S198785. eCollection 2020. PMID 32754451
- [Background] Young NA, Sharma M, Deogaonkar M. Transcranial magnetic stimulation for chronic pain. Neurosurg Clin N Am. 2014 Oct;25(4):819-32. doi: 10.1016/j.nec.2014.07.007. Epub 2014 Aug 12. PMID 25240669
- [Background] Ziegelmann MJ, Farrell MR, Levine LA. Evaluation and Management of Chronic Scrotal Content Pain-A Common Yet Poorly Understood Condition. Rev Urol. 2019;21(2-3):74-84. PMID 31768134